CLINICAL TRIAL: NCT06334471
Title: Whole Genome Sequencing in Breast Cancer
Acronym: WGS SIT
Status: Recruiting | Type: Observational
Sponsor: Inocras Korea Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: INCS_WGS_B-001
Record Dates: First submitted 2024-03-20; First posted 2024-03-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; whole genome sequencing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — In both prospective and retrospective studies, individual identifiers for each research subject and specimen are anonymized, and research subject numbers are assigned to manage the specimens. Specimens collected in the prospective study of this research will be identified by coded numbers, and their retention and disposal will be determined based on the specified retention period in the informed consent form, provision availability for other research purposes, and procedures for handling personal information upon provision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prospective study: The prospective study group includes patients aged 19 years or older who have provided written consent for participation, have the capability to consent voluntarily, are eligible for tissue examination and surgical removal for sample collection, and have confirmed or suspected breast cancer for pathological confirmation.
  Interventions: Other: no intervention needed
- Retrospective study: The retrospective study group includes patients who have been histologically confirmed with breast cancer and whose breast cancer tissues collected between 2012 and 2023 are stored in the Samsung Seoul Hospital Human Biobank and available for distribution.
  Interventions: Other: no intervention needed

INTERVENTIONS:
Other: no intervention needed — no intervention needed

SUMMARY:
This study aims to conduct whole genome sequencing in breast cancer patients to elucidate individual genetic characteristics and their correlation with breast cancer subtypes. The primary objective is to establish new treatment guidelines aligned with the paradigm shift in precision medicine. The study will include both prospective and retrospective cohorts totaling 1200 participants. Prospective participants must provide consent and be eligible for tissue collection, while retrospective participants must have histologically confirmed breast cancer and available tissue samples from Samsung Medical Center Biobank. The study period spans 3 years for subject enrollment and 5 years for follow-up observations, with an expected completion date of December 31, 2030.

DETAILED DESCRIPTION:
Breast cancer is a complex disease with diverse genetic characteristics, necessitating personalized treatment approaches. This study proposes to conduct whole genome sequencing (WGS) to comprehensively analyze the genetic landscape of breast cancer patients, aiming to identify novel genetic alterations and their implications for disease classification and treatment response.

The primary objective of this research is to elucidate the individual genetic profiles of breast cancer patients through WGS and subsequent analysis. By characterizing the genomic alterations unique to each patient, this study seeks to refine breast cancer subtyping, facilitate the discovery of innovative treatment strategies, and optimize therapeutic decision-making.

This multicenter study will enroll a total of 1200 participants, comprising both prospective and retrospective cohorts. Prospective participants will be recruited based on specific inclusion criteria, including age, consent for tissue collection, and histologically confirmed breast cancer diagnosis. Retrospective participants will be identified from existing breast cancer tissue samples collected between 2012 and 2023 and stored in the Samsung Medical Center Biobank.

The study will involve comprehensive data collection, including clinical, pathological, and genomic information. Participants will undergo WGS analysis of tumor samples, and the resulting genomic data will be correlated with clinical outcomes to identify potential prognostic markers and therapeutic targets.

The research will be conducted under the supervision of Professor Yeonhee Park, an expert in hematology-oncology at Samsung Medical Center, in collaboration with Inocras Inc, the study sponsor. The study period will span three years for subject enrollment, followed by a five-year follow-up observation period. The expected completion date for the study is December 31, 2030.

This study holds the potential to significantly advance our understanding of the molecular basis of breast cancer and pave the way for the development of personalized treatment approaches tailored to individual patients' genetic profiles.

ELIGIBILITY:
[Prospective study]

Inclusion Criteria:

* Patients who have consented to both the patient consent form and the consent for the use of human-derived materials.
* Patients who are aged 19 years or older at the time of signing the consent form.
* Patients capable of providing written consent to participate voluntarily in the study.
* Patients eligible for tissue examination and surgical removal to facilitate sample collection.
* Patients histologically confirmed with breast cancer or undergoing tissue examination for pathological confirmation due to imaging findings suggestive of breast cancer.

Exclusion Criteria:

* Patients who do not understand or refuse to consent in writing.
* Patients for whom obtaining sufficient samples is challenging.
* Patients who refuse genetic testing.

[Retrospective study]

Inclusion Criteria:

* Patients histologically confirmed with breast cancer.
* Patients for whom breast cancer tissues collected between 2012 and 2023 are stored in the Samsung Seoul Hospital Biobank and available for distribution.

Exclusion Criteria:

- Patients for whom sufficient tissue for analysis is not adequately stored.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prospective study : 500 Retrospective study : 700
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-08-02 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Establishing individual genetic characteristics of breast cancer patients through WGS | December.31.2030
  The primary goal of this study is to elucidate the individual genetic traits of breast cancer patients through comprehensive analysis of their whole genome and observational factors.

SECONDARY OUTCOMES:
Analysis of correlation between whole-genome sequencing results and genetic subtypes of breast cancer | December.31.2030
  Analysis of correlation between whole-genome sequencing results and genetic subtypes of breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: JeongSeok Lee, Study Chair — Inocras Korea Inc.
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No